## **Informed Consent Form**

Small/diminutive polyp training module using novel endoscopic imaging: a comparison between didactic training and self-directed computer based training

| I | D: | / | | |
|---|---|---|---|---|
| I | nitials: | | | |
| P | rincipal Investigator: | | | |
| | | | Please initial inside eac | ch box |
| 1 | I confirm that I have read and understood the information sheet, dated $\_\_/\_\_/$ version number $\_\_$ . $\_\_$ for the <i>polyp training module</i> . I have had the opportunity to consider the information, ask questions, and have had these answered satisfactorily. | | | |
| 2 | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason. I understand that data collected up to my time of withdrawal may be used. | | | |
| 3 | I understand data collected from me during the study will be looked at by individuals from the research team, representatives of the sponsor, from regulatory authorities, or from the NHS Trust, where this is relevant. I give permission for these individuals to have direct access to the data I supply. | | | |
| 5 | Data collected that identifies me by name, (consent form and registration forms), will be transferred from where it is collected and stored at the University of Birmingham, I agree to the transfer and storage of this data. | | | |
| 6 | I understand that the information I have given you will be stored at the University of Birmingham, and that this data will be destroyed when it is no longer needed in accordance with the Data Protection Act 1988. I agree to this data being stored. | | | |
| 7 | I agree to take part in this st | audy. | | |
| | lame of Participant | | <br>Signature | |
| | , | | <b>5</b> | |